CLINICAL TRIAL: NCT02022436
Title: Aortic Wall Behavior as a Predictor of Aortic Aneurysm Growth and Rupture
Brief Title: Evaluation of Predictors of Aortic Aneurysm Growth and Rupture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabih A. Chaer (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Rabih A. Chaer, Associate Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AG042352-01; 1R03AG042352-01 (NIH)
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- contrast ultrasound for patients with AAA (Active Comparator): Contrast ultrasound
  Interventions: Drug: Contrast Ultrasound
- contrast ultrasound for patients without arterial disease (Active Comparator): contrast enhanced ultrasound
  Interventions: Drug: Contrast Ultrasound

INTERVENTIONS:
Drug: Contrast Ultrasound — Definity® is the contrast agent that will be administered by intravenous injection by a registered nurse during the ultrasound (contrast enhanced ultrasound (CUS). The purpose is to assist in identifying differences in AAA characteristics based on gender and AAA stability and growth.
  Other Names: Definity

SUMMARY:
The goal is to non-invasively study the metabolic processes within the aortic wall that are thought to explain progression to clinical manifestations of an aortic aneurysm.

Hypothesis is that the non-invasive imaging of Abdominal Aortic Aneurysm (AAA) with contrast ultrasound, coupled with serum biomarker measurements will allow the identification of the vulnerable aortic wall and patients who are at risk of AAA growth or rupture.

DETAILED DESCRIPTION:
Aim#1: Prospective Contrast Ultrasound (CUS) imaging of patients with AAA to predict AAA growth and test gender differences in rate of growth and rupture.

Aim#2: Serum biomarker testing of patient with AAA. CUS findings will be correlated with serum biomarkers and AAA wall histology.

Prospective Contrast Ultrasound imaging of patients with AAA as part of a pilot feasibility study to predict AAA growth and test gender differences in rate of growth and rupture. CUS findings will be correlated with serum biomarkers and AAA wall histology. Potential significance: This study will evaluate the AAA wall and will be based on detecting areas of increased vasa vasorum density within the aneurysm wall and intraluminal thrombus, which indicate regional ischemia and inflammation of the aortic wall and propensity for weakening, enlargement or rupture. This novel evaluation of the aortic wall in patients with AAA will allow individualized treatment based on the biological potential for growth and rupture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AAA with confirmation of diagnosis of any size aneurysm with imaging.
* 21 years of age or older
* ability to give informed consent.

Exclusion Criteria:

* Inability to provide an informed consent
* Known allergy to Definity
* Unstable cardiopulmonary conditions
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Chaer, MD, Principal Investigator — UPMC UPP
Locations (1):
- University of Pittsburgh Medical Center, Division of Vascular Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast Ultrasound for Patients With AAA | Contrast Ultrasound for Patients Without Arterial Disease
Started | 59 | 7
Completed | 59 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contrast Ultrasound for Patients With AAA | Contrast Ultrasound for Patients Without Arterial Disease | Total
Number analyzed (Participants) | 59 | 7 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 6 | 24
  >=65 years | 41 | 1 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (8.6) | 49.4 (12.8) | 67.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 51 | 1 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 55 | 4 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 59 | 7 | 66

OUTCOME MEASURES:

1. Primary Outcome: Annual Aneurysm Growth Rate Between Patients With and Without Micro Bubble Uptake
Description: Prospective contrast ultrasound will be performed at regular clinically indicated timepoints.
Time Frame: Up to 5 years or time of aneurysm repair surgery.
Population: Annual aneurysm growth rate only relevant for patients with aneurysm disease
Measure: Mean (Standard Deviation); unit: mm/year
Groups:
- Contrast Ultrasound for Patients With Aneurysm Disease: Contrast ultrasound
  contrast ultrasound: Definity® is the contrast agent that will be administered by intravenous injection by a registered nurse during the ultrasound (contrast enhanced ultrasound (CUS). The purpose is to assist in identifying differences in AAA characteristics based on gender and AAA stability and growth.
  Contrast Ultrasound: Definity® is the contrast agent that will be administered by intravenous injection by a registered nurse during the ultrasound (contrast enhanced ultrasound (CUS). The purpose is to assist in identifying differences in AAA characteristics based on gender and AAA stability and growth.
Arm/Group | Contrast Ultrasound for Patients With Aneurysm Disease
Number analyzed (Participants) | 59
mm/year
  Microbubble Uptake: number analyzed (Participants) | 36
  Microbubble Uptake | 3.0 (3.1)
  No Microbubble Uptake: number analyzed (Participants) | 23
  No Microbubble Uptake | 3.2 (3.1)

2. Primary Outcome: Number of Participants With Microbubble Uptake
Description: Microbubble uptake was determined on ultrasound evaluation of the abdominal aorta. This was agreed upon by two reading physicians.
Time Frame: At the first follow-up evaluation at 6 months
Population: Microbubble Uptake was only evaluated in patients with aneurysm disease as patients without aneurysm disease do not have micro bubble uptake.
Measure: Count of Participants; unit: Participants
Groups:
- Contrast Ultrasound for Patients With AAA: Contrast ultrasound contrast ultrasound: Definity® is the contrast agent that will be administered by intravenous injection by a registered nurse during the ultrasound (contrast enhanced ultrasound (CUS). The purpose is to assist in identifying differences in AAA characteristics based on gender and AAA stability and growth.
  Contrast Ultrasound: Definity® is the contrast agent that will be administered by intravenous injection by a registered nurse during the ultrasound (contrast enhanced ultrasound (CUS). The purpose is to assist in identifying differences in AAA characteristics based on gender and AAA stability and growth.
Arm/Group | Contrast Ultrasound for Patients With AAA
Number analyzed (Participants) | 59
Participants | 36

3. Secondary Outcome: Mean Value of Systemic Inflammatory Serum Biomarkers
Description: Systemic serum biomarkers of AAA will be measured. These markers are circulating levels of C Reactive Protein, cytokines and osteoprotegerin.
  Serum markers will be drawn at baseline and at the next follow-up visit which is 6 months after the index visit.
Time Frame: baseline, 6 months
Population: For patients without arterial disease, serum biomarkers were only obtained at baseline; no follow-up visits occurred and therefore no further biomarker testing was done.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Contrast Ultrasound for Patients With AAA | Contrast Ultrasound for Patients Without Arterial Disease
Number analyzed (Participants) | 59 | 7
pg/ml
  Osteoprotegrin | 225.5 [142.7 to 308.3] | 214.8 [134.7 to 294.9]
  C Reactive Protein | 7090.3 [3619.0 to 10561.6] | 1843.0 [1017.2 to 2668.8]
  Interferon | 4.2 [3.3 to 4.8] | 2.4 [1.8 to 2.9]
  Osteoprotegrin (at 6 months): number analyzed (Participants) | 59 | 0
  Osteoprotegrin (at 6 months) | 257.4 [225.0 to 289.8] |
  C Reactive Protein (at 6 months): number analyzed (Participants) | 59 | 0
  C Reactive Protein (at 6 months) | 7808.0 [220.2 to 15395.8] |
  Interferon (at 6 months): number analyzed (Participants) | 59 | 0
  Interferon (at 6 months) | 5.1 [3.5 to 6.6] |

ADVERSE EVENTS:
Time Frame: Adverse data were collected from the time of contrast administration through study completion (an average of 6 months), for all patients.
Description: The definitions do not differ.
Arm/Group | Contrast Ultrasound for Patients With AAA | Contrast Ultrasound for Patients Without Arterial Disease
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/7
Other Adverse Events (participants affected / at risk) | 0/59 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02022436/Prot_SAP_000.pdf